CLINICAL TRIAL: NCT01541891
Title: Fase II Comparative Study of the Efficacy and Safety of PRO-148 Ophthalmic Solution vs Systane in the Treatment of Mild-to-moderate Eye Syndrome.
Brief Title: Efficacy and Safety of PRO-148 Ophthalmic Solution Versus SYSTANE® in the Treatment of Patients With Dry Eye Syndrome
Acronym: PRO-148
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COXAVSSY0311FII; PRO-148 (Other: SOPHIA PRO-148)
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-02

CONDITIONS: Dry Eye Syndrome
Keywords: PRO-148; Dry eye syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO-148 Ophthalmic Solution (Experimental): Drug: PRO-148 Intervention name: PRO-148 applied in ocular surface of patients with mild to moderate dry eye syndrome q.i.d. for 60 days
  Interventions: Drug: PRO-148 Ophthalmic Solution
- Arm B. SYSTANE® Ophthalmic Solution (Active Comparator): Drug: SYSTANE® Intervention name: SYSTANE® applied in ocular surface of patients with mild to moderate dry eye syndrome q.i.d. for 60 days
  Interventions: Drug: Active Comparator: SYSTANE ® Ophthalmic Solution

INTERVENTIONS:
Drug: PRO-148 Ophthalmic Solution — PRO-148 Ophthalmic Solution applied four times per day (c/6 hours) during 60 days.
  Other Names: PRO-148
  Arms: PRO-148 Ophthalmic Solution
Drug: Active Comparator: SYSTANE ® Ophthalmic Solution — Sterile solution containing polyethylene glycol 400, propylene glycol, hydroxypropyl-guar, boric acid, calcium chloride, magnesium chloride, potassium chloride, sodium chloride, zinc chloride and polyquad (polidronium chloride) 0,001%. four times per day (c/6 hours) during 60 days.
  Arms: Arm B. SYSTANE® Ophthalmic Solution

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PRO-148 ophthalmic solution compared with SYSTANE ® ophthalmic solution for the treatment of signs and symptoms of mild-to-moderate dry eye syndrome.

DETAILED DESCRIPTION:
A phase 2, randomized, double masked clinical, parallel-group clinical trial to evaluate the efficacy and safety of PRO-148 ophthalmic solution compared with SYSTANE ® ophthalmic solution for the treatment of signs and symptoms of mild-to-moderate dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of mild-to-moderate drye eye syndrome.
* Male or female patients.
* Patients 18 years of age

Exclusion Criteria:

* Patients with one blind eye.
* Visual acuity of 20/40 in any eye
* Patients with history of active stage of any other concomitant ocular disease.
* Patients taking any medication, topically or by any other route, which could interfere with the study's results, in the 3 days prior to trial or until a time period in which residual effects could be present.
* Contraindications or sensitivity to any component of the study treatments.
* Ocular surgery within the past 3 months.
* Contact lens users.
* Females of childbearing potential )may not participate in the study if any of the following conditions exist:

  * They are pregnant,
  * They are breastfeeding,
  * They have a positive urine pregnancy test at screening,
  * They intend to become pregnant during the study, or
  * They do not agree to use adequate birth control methods for the duration of the study.
* Participation in any studies of investigational drugs within 90 days previous to the inclusion.

Discontinuation criteria:

* Patients could be discontinued before the completion of the study because of adverse events, pregnancy, protocol violations, lack of efficacy, or administrative reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José F Alaniz-De La O, MD, Principal Investigator — Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde"; Laura R Saucedo-Rodíguez, MD, Principal Investigator — Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde"; Leopoldo M Baiza-Durán, MD, Study Director — Clinical Research Department. Laboratorios Sophia SA de CV
Locations (1):
- Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were enrolled in this study at 1 hospital
Pre-assignment Details: Elegible patients were de novo patients diagnosed with mild to moderate dry eye disease
Groups:
- Arm A PRO 148 Ophthalmic Solution: PRO-148 Ophthalmic Solution : PRO-148 Ophthalmic Solution applied four times per day (c/6 hours) during 60 days.
- Arm B. SYSTANE® Ophthalmic Solution: Active Comparator: SYSTANE ® Ophthalmic Solution : Sterile solution containing polyethylene glycol 400, propylene glycol, hydroxypropyl-guar, boric acid, calcium chloride, magnesium chloride, potassium chloride, sodium chloride, zinc chloride and polyquad (polidronium chloride) 0,001%. four times per day (c/6 hours) during 60 days.
Period: Overall Study
Arm/Group | Arm A PRO 148 Ophthalmic Solution | Arm B. SYSTANE® Ophthalmic Solution
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 14 patients of each group were included in the analysis (28 i total), the other 2 patients (1 of each group) were excluded due to lack of follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A PRO 148 Ophthalmic Solution | Arm B. SYSTANE® Ophthalmic Solution | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (8.4) | 55.9 (9.6) | 55.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Mexico | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Break-up Time (TBUT)
Description: TBUT was evaluated at baseline and end of the study
Time Frame: During 60 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arm A PRO 148 Ophthalmic Solution | Arm B. SYSTANE® Ophthalmic Solution
Number analyzed (Participants) | 14 | 14
seconds
  Baseline | 5.2 (2.3) | 4.7 (2.6)
  End of the study | 6.1 (2.5) | 7.3 (2.5)

2. Secondary Outcome: Presence of Adverse Events
Description: The presence of adverse events will be reported in both treatment arms. This variable will be reported by the number of events presented.
Time Frame: 60 days
Measure: Number; unit: number of cases
Arm/Group | Arm A PRO 148 Ophthalmic Solution | Arm B. SYSTANE® Ophthalmic Solution
Number analyzed (Participants) | 14 | 14
number of cases | 1 | 0

3. Other Pre Specified Outcome: Evaluation of Visual Acuity
Description: The LogMAR scale evaluates the visual acuity of subjects with a logarithmic scale where base 0 is the best visual acuity and 1 is the worst. This variable will be reported with means for comparison between groups.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on LogMAR scale
Groups:
- PRO-148: Drug: PRO-148 Intervention name: PRO-148 applied in ocular surface of patients with mild to moderate dry eye syndrome
  PRO-148 Ophthalmic Solution: PRO-148 Ophthalmic Solution applied four times per day (c/6 hours) during 60 days.
Arm/Group | PRO-148 | Arm B. SYSTANE® Ophthalmic Solution
Number analyzed (Participants) | 14 | 14
units on LogMAR scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Arm A PRO 148 Ophthalmic Solution | Arm B. SYSTANE® Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A PRO 148 Ophthalmic Solution (N=14) | Arm B. SYSTANE® Ophthalmic Solution (N=14)
Cephalea (Investigations) | 1 | 0 — An adverse event was present (mild-intensity cephalea at visit 1 that did not need medications for its relief) in the CS/XG group, but it was not related to the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information is confidential and exclusive property of the sponsor. Information can be revealed only to my staff and regulatory agencies or ethics committee.

All the information from this protocol is confidential and exclusive property of the sponsor, it can not be revealed without written consent from the sponsor.